CLINICAL TRIAL: NCT07363499
Title: Combining Physical Activity and Sedentary Interventions to Improve Cardiometabolic Health
Acronym: CAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Prof Dr. Bert Op 't Eijnde, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CME2024/069
Record Dates: First submitted 2025-12-22; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cardiometabolic Risk Factors; Sedentary Behaviors; Insulin Resistance
Keywords: Cardiometabolic health; Sedentary behaviour; Physical activity; Exercise; Insulin resistance
MeSH Terms: conditions — Sedentary Behavior; Insulin Resistance; Motor Activity

STUDY DESIGN:
Intervention Model Description: First all participants will follow a control period after which they are randomised to a parallel design with two intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (2 weeks) (No Intervention): All participants will follow a two-week period where no intervention is administered.
- PA group (8 weeks) (Active Comparator): After the control period without intervention, one halve of the participants is randomised to the PA group where participants are encouraged to adhere to WHO physical activity guidelines during 8 weeks.
  Interventions: Behavioral: WHO physical activity guideline
- PA-SB group (8 weeks) (Experimental): After the control period without intervention, one halve of the participants is randomised to the PA-SB group where participants are encouraged to adhere to WHO physical activity guidelines. In addition, sedentary time at the workplace is reduced. The duration of this intervention is 8 weeks.
  Interventions: Behavioral: WHO physical activity guideline; Behavioral: Sedentary behaviour reduction at the workplace

INTERVENTIONS:
Behavioral: WHO physical activity guideline — Individualised Physical Activity Plan (8 weeks):
  • Two weekly sessions of moderate-intensity physical activity (MIPA): Frequency: 2 sessions per week. Unsupervised. Duration: Initially 40 minutes per session, increasing to 50 minutes by week 4. Type of Activity: Participants can select from brisk walking, cycling, swimming, or elliptical training.
  Intensity: 40-60% of maximal oxygen consumption, monitored with wearable heart rate devices.
  • One weekly session of vigorous-intensity physical activity (VIPA): Frequency: 1 session per week. Supervised or predetermined. Duration: Initially 20 minutes per session, increasing to 30 minutes by week 4. Type of Activity: Options include running, high-intensity interval training (HIIT), or fast cycling.
  Intensity: 60-90% of maximal oxygen consumption, tracked with heart rate devices.
  • Weekly check-ins will allow adjustments based on individual feedback and progress.
  Arms: PA group (8 weeks); PA-SB group (8 weeks)
Behavioral: Sedentary behaviour reduction at the workplace — Participants will be encouraged to replace seated work with standing work and engage in light physical activity breaks.
  • Workplace Integration Strategies: Participants working in an office setting will be provided with adjustable sit-stand desks where possible.
  • Active Breaks and Movement Interventions: Participants will be prompted to take short (2min) active breaks after prolonged periods of sedentary behaviour.
  Break activities will include standing, stretching, or light movement such as walking.
  Arms: PA-SB group (8 weeks)

SUMMARY:
Many adults spend a large part of their day sitting, especially at work. Long periods of sitting and not moving enough can increase the risk of health problems such as heart disease and type 2 diabetes. This risk is even higher in people who have early warning signs like being overweight, having high blood pressure, or problems with blood sugar. Together, these problems are called metabolic syndrome.

The goal of this study is to find out whether combining regular exercise with reducing sitting time during the day can improve heart and metabolic health more than exercise alone.

About 40 adults between 18 and 65 years old who work mainly at a desk and sit for more than 9 hours a day will take part. All participants will first continue their normal daily routine for two weeks. After that, they will be randomly placed into one of two groups for eight weeks:

Exercise group: Participants will follow the World Health Organization guidelines for physical activity. This includes two sessions of moderate exercise each week (such as brisk walking or cycling) and one session of more intense exercise each week.

Exercise plus less sitting group: Participants will do the same exercise program, but they will also be encouraged to sit less during the workday. They will be asked to stand more, use sit-stand desks if possible, and avoid sitting for longer than one hour at a time.

Participants will visit the research center three times for health tests. These tests include blood samples to look at blood sugar, insulin, and fats in the blood, measurements of blood pressure and heart function, body composition scans, fitness tests, and questionnaires about sleep, diet, and quality of life. They will also wear activity monitors to measure how much they sit, stand, and move.

The main outcome is how the body handles sugar (insulin sensitivity). The researchers hope to learn whether sitting less, in addition to exercising, leads to better improvements in heart and metabolic health. The results may help develop better lifestyle advice to prevent heart disease and diabetes in people with desk jobs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Profession where most of the time is spent sitting.
* Not regularly physically active (>3 trainings per week in the last three months)
* Sedentary (on average >9 hours per day spent sedentary on a working day)
* Written informed consent to participate in the study.

Exclusion Criteria:

* Pregnancy.
* Consumption of more than 20 units of alcohol per week.
* Medical conditions that limit physical activity.
* Specific diet (e.g. low-carbohydrate or calorie-restricted).
* Unstable body weight in the past month.
* Participation in another study that could potentially affect your blood parameters in the past month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Homeostatic model assessment for insulin resistance (HOMA-IR) | From enrollment to the end of the intervention at 8 weeks.
  The HOMA-IR is calculated from the fasting insulin and glucose concentration.
Whole-body insulin sensitivity index (ISI) | From enrollment to the end of the intervention at 8 weeks
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity using the whole-body insulin sensitivity index (ISI). The ISI is calculated from both insulin and glucose concentrations.
Area under the curve of insulin concentrations | From enrollment to the end of the intervention at 8 weeks
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity by calculation of the area under the curve of insulin concentrations.
Insulinogenic index | From enrollment to the end of the intervention at 8 weeks.
  An oral glucose tolerance test will be performed for assessment of beta cell function by calculation of the insulinogenic index. The insulinogenic index is calculated from both insulin and glucose concentrations.

SECONDARY OUTCOMES:
Body composition | From enrollment to the end of the intervention at 8 weeks.
  Body composition is evaluated by Dual-energy X-ray absorptiometry. Fat mass (in kg), lean body mass (in kg), body fat percentage (in %) and visceral adipose tissue (in grams) will be derived from the Dual-energy X-ray absorptiometry.
Cardiorespiratory Fitness | From enrollment to the end of the intervention at 8 weeks.
  Cardiorespiratory fitness will be measured as peak oxygen consumption (V̇O2peak) using a graded cardiopulmonary exercise test (CPET) on a bike with pulmonary gas exchange analysis (Jaeger Oxycon®) until volitional exhaustion.
Area under the curve of glucose concentrations | From enrollment to the end of the intervention at 8 weeks
  An oral glucose tolerance test will be performed for assessment of whole body insulin sensitivity by calculation of the area under the curve of glucose concentrations.
Steps per day | From enrollment to the end of the intervention at 8 weeks. For one week during the first four weeks of the intervention. For one week during the last four weeks of the intervention.
  Physical activity will be quantified using the activPAL3™ activity monitor.
Sitting time | From enrollment to the end of the intervention at 8 weeks. For one week during the first four weeks of the intervention. For one week during the last four weeks of the intervention.
  Sedentary behaviour will be quantified using the activPAL3™ activity monitor.
Moderate to vigorous physical activity | From enrollment to the end of the intervention at 8 weeks. For one week during the first four weeks of the intervention. For one week during the last four weeks of the intervention.
  Physical activity will be quantified using the activPAL3™ activity monitor.
Light intensity physical activity | From enrollment to the end of the intervention at 8 weeks. For one week during the first four weeks of the intervention. For one week during the last four weeks of the intervention.
  Physical activity will be quantified using the activPAL3™ activity monitor.
Sleep | From enrollment to the end of the intervention at 8 weeks. For one week during the first four weeks of the intervention. For one week during the last four weeks of the intervention.
  Physical activity will be quantified using the activPAL3™ activity monitor.
Body weight | From enrollment to the end of the intervention at 8 weeks
  Body weight (in underwear) is determined using a digital-balanced weighting scale to the nearest 0.1kg
Height | From enrollment to the end of the intervention at 8 weeks.
  Body height is measured to the nearest 0.1cm using a wall-mounted Harpenden stadiometer, with participants barefoot
Body mass index | From enrollment to the end of the intervention at 8 weeks
  Body mass index (BMI; kg/m²) is calculated from weight and height measurements (weight/height²).
Waist and hip circumference | From enrollment to the end of the intervention at 8 weeks
  Waist and hip circumferences will be measured to the nearest 0.1 cm using a flexible metric measuring tape with participants barefoot (in underwear) in standing position. Waist circumference is measured at the midpoint between the lower rib margin and the top of the iliac crest. Hip circumference is measured at the widest circumference of the hip at the level of the greater trochanter. Waist-to-hip ratio is calculated by dividing waist circumference (cm) by hip circumference (cm). Waist-to-height ratio is calculated by dividing waist circumference (cm) by height (cm).
Blood pressure | From enrollment to the end of the intervention at 8 weeks
  After an initial resting period of 10 min with participants in a supine position in a quiet room with constant temperature (21°C), systolic and diastolic blood pressure (BP; in mmHg) will be measured at least 3 times at 2-min intervals until BP is stable using an electronic sphygmomanometer (Omron®) from the left arm and documented as the mean value of the three final measurements.
Vascular endothelial function | From enrollment to the end of the intervention at 8 weeks
  Vascular function will be assessed by FMD according to published guidelines. These measurements take place at 9h and involve doppler ultrasound imaging of the superficial femoral artery. A cuff will be placed on the right lower leg, and the superficial femoral artery is imaged longitudinally. FMD will be measured at baseline and after a 5-min occlusion phase (reactive hyperaemia response). FMD will be quantified as the percentage difference between peak and baseline diameter (FMD%).
Cardiac autonomic function | From enrollment to the end of the intervention at 8 weeks
  Cardiac autonomic function will be operationalized as heart rate variability by means of continuous beat-to-beat heart rate signal measurements. time domain and frequency domain analysis of the R-R intervals will be performed
Concentration of glucose | From enrollment to the end of the intervention at 8 weeks
  Blood analysis
Concentration of insulin | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of total cholesterol | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of Low-Density Lipoprotein cholesterol | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of High-Density Lipoprotein cholesterol | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of triglycerides | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of apolipoproteins | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of CRP | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of Interleukin 6 (IL-6) | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Concentration of interleukin 1 (IL-1) | From enrollment to the end of the intervention at 8 weeks.
  Blood analysis
Sleep quality | From enrollment to the end of the intervention at 8 weeks.
  Sleep quality over a period of one month will be assessed with the Pittsburgh sleep quality index (PSQI) which is a self-administered questionnaire consisting of 19 items that is reliable and valid to assess sleep problems.
Food intake | From enrollment to the end of the intervention at 8 weeks
  Habitual dietary intake is assessed using a validated food frequency questionnaire (FFQ). In addition, participants will fill in a diary to evaluate dietary intake either with an app or on paper.
Quality of life (QOL) | From enrollment to the end of the intervention at 8 weeks
  Health-related quality of life (HRQOL) was measured using the Euroqol 5-D questionnaire (EQ-5D). The EQ-5D is a widely used and validated generic instrument consisting of five dimensions: mobility, self- care, usual activities, pain/discomfort and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jen Vanherle, MSc, Principal Investigator — Hasselt University
Locations (1):
- Univeristeit Hasselt, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
In a restriced access depositry. Personal data is sensitive data and is thus protected in a restricted access repository. During the project these data will be pseudonymized and after completion of the project data will be anonymized and the pseudonymization key will be destroyed. Access can be granted by the primary investigator who holds the pseudonymization key in a restricted folder during the project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the results, data will become available for a duration of 25 years.
Access Criteria: Access will be granted after motivated and reasonable request to the principal investigator.